CLINICAL TRIAL: NCT07058831
Title: Home Monitoring for the Detection of Subclinical Atrial Fibrillation in Hypertensive Patients at Moderate to High Risk of Developing Arrhythmia. BP/AF MODE Study.
Brief Title: Subclinical Atrial Fibrillation Home Monitoring in Hypertensive Patients
Status: Recruiting | Type: Observational
Sponsor: Cardiovascular Research Center Rosario British Sanatorium (Other)
Responsible Party: Principal Investigator, Daniel L Piskorz, Director, Cardiovascular Research Center Rosario British Sanatorium
Other Study IDs: PA/AF Mode
Record Dates: First submitted 2025-06-24; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Asymptomatic Atrial Fibrillation
Keywords: hypertension; atrial fibrillation; home monitoring; artificial intelligence
MeSH Terms: conditions — Hypertension; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Hypertensive patients older 75 or Hypertensive patients between 65 and 75 at moderate-high risk AF: The 30-second home ECG tracings will be obtained using the Omron Complete Hem-7530 T ECG device (Omron Healthcare Co., Ltd., Japan). The connection and smartphone app download will be available from Omron Connect free of charge on the Google Play Store: https://play.google.com/store/apps/details?id=jp.co.omron.healthcare.omron_connect&hl=es_419&pli=1 and on the iOS App Store: https://apps.apple.com/mx/app/omron-connect/id1003177043. Two duplicate ECG recordings will be required daily: the first in the morning before breakfast and taking the prescribed medication, and another in the evening before dinner and taking the afternoon/evening medication. Additional ECG recordings will be required if the patient experiences any symptoms.
  Interventions: Device: Home ECG monitoring

INTERVENTIONS:
Device: Home ECG monitoring — The 30-second home ECG tracings will be obtained using the Omron Complete Hem-7530 T ECG device (Omron Healthcare Co., Ltd., Japan). The connection and smartphone app download will be available from Omron Connect free of charge on the Google Play Store: https://play.google.com/store/apps/details?id=jp.co.omron.healthcare.omron_connect&hl=es_419&pli=1 and on the iOS App Store: https://apps.apple.com/mx/app/omron-connect/id1003177043. Two duplicate ECG recordings will be required daily: the first in the morning before breakfast and taking the prescribed medication, and another in the evening before dinner and taking the afternoon/evening medication. Additional ECG recordings will be required if the patient experiences any symptoms.

SUMMARY:
Atrial fibrillation is a highly prevalent and incidental arrhythmia, often asymptomatic, and frequently detected incidentally or in association with a stroke. Subclinical atrial fibrillation increases cardioembolic risk, highlighting the need for timely diagnosis.

New wireless devices capable of recording heart rhythm, combined with innovative artificial intelligence tools, could be useful in the prediction and detection of this arrhythmia.

Objective: to determine the usefulness of home blood pressure and heart rhythm monitoring strategy in the detection of subclinical atrial fibrillation.

Methods: observational, cohort, prospective, multicenter study involving 25 researchers from six Latin American countries. Home blood pressure monitoring and single-lead electrocardiogram recording were performed in a population at moderate to high risk of developing atrial fibrillation. A minimum of twenty 30-second electrocardiographic and blood pressure recordings over 7 days using an Omron Complete Hem-7530 T ECG device will be uploaded from a mobile phone app and then sent to a database for analysis.

Conclusions: the results of this study can provide a simple and accessible home monitoring system for detecting subclinical atrial fibrillation and for optimizing the predictive capacity of arrhythmia risk scores through deep learning.

DETAILED DESCRIPTION:
The BP/AF Mode study is a multicenter, observational, prospective, cohort trial involving 25 researchers from six countries: Argentina, Chile, Colombia, Ecuador, Mexico, and Peru. The study was submitted to the IASC Academia (Inter-American Society of Cardiology) and approved under Project File Number 052, dated January 29, 2025. It will be conducted in full compliance with the World Medical Association Codes of Ethics for experiments involving human subjects.

The study aims to include hypertensive patients with no history of atrial fibrillation who are at moderate or high risk of suffering from this arrhythmia according to the HARMS2-AF score or the modified Taiwan AF . The diagnosis of hypertension is supported on the 2023 European Society of Hypertension Guidelines. The patients' baseline characteristics are entered into an interactive web platform, and after that the practitioners received information about cardiovascular risk (Hearts score, Score-2 and Score-OP), Frailty index and atrial fibrillation risk (HARMS2-AF score and modified Taiwan AF score).

After the screening visit, if the patient meets all the inclusion criteria and does not present exclusion criteria, he or she is included in the study and a Omron Complete Hem-7530 T ECG device (Omron Healthcare Co., Ltd., Japan) device is delivered.

The 30-second home ECG tracings will be obtained using the Omron Complete Hem-7530 T ECG device (Omron Healthcare Co., Ltd., Japan). The connection and smartphone app download will be available from Omron Connect free of charge on the Google Play Store: https://play.google.com/store/apps/details?id=jp.co.omron.healthcare.omron_connect&hl=es_419&pli=1 and on the iOS App Store: https://apps.apple.com/mx/app/omron-connect/id1003177043. Two duplicate ECG recordings will be required daily: the first in the morning before breakfast and taking the prescribed medication, and another in the evening before dinner and taking the afternoon/evening medication. Additional ECG recordings will be required if the patient experiences any symptoms. The study investigator will work with the patient to download the app and perform the first electrocardiogram tracing and transmit it to the database. The patient will be given instructions on how to correctly perform the ECG and transmit it to the platform, along with a patient diary. Simultaneously with obtaining the ECG tracings, the patient will take two BP measurements, in a seated position, separated by one minute, following the recommendations of the Latin American Society of Hypertension guidelines. After 1 week, the patient will return the device to the research center. A recording will be considered valid when at least 80% of the ECG tracings and BP measurements are valid.

Statistical analysis Considering those patients with a modified Taiwan AF score > 5 points, whose annual incidence of atrial fibrillation ranges between 1.54% and 6.98%, or a HARMS2-AF score > 7 points, whose annual incidence of atrial fibrillation ranges between 1.35% and 6.62%, it will be required to include 499 patients to achieve a 5% margin of error, with a 99% confidence level. If the sample calculation does not achieve the expected results, recruitment will continue until 25 cases of atrial fibrillation are reached.

Continuous variables will be reported as means with their standard deviations for normally distributed variables, or median and interquartile range for non-normally distributed variables. Discrete variables will be reported as absolute values and percentages. Unpaired ANOVA will be used to analyze normally distributed variables, while the Kruskal-Wallis test will be used for non-normally distributed variables. Differences in proportions will be assessed using the Chi-square test. A two-tailed p-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1. Hypertensive patients of both sexes over 75 years of age. 2. Hypertensive patients between 65 and 75 years of age are associated with one of the following risk factors:

  1. Obesity
  2. Type 2 diabetes
  3. Obstructive sleep apnea syndrome
  4. Electrocardiogram showing left ventricular hypertrophy.
  5. Left ventricular hypertrophy on echocardiogram.
  6. Left atrial dilation.
  7. Coronary artery disease
  8. Chronic kidney disease
  9. Heart failure with ejection fraction > 50%
  10. Alcohol intake
  11. Frequent supraventricular ectopic beats

Exclusion Criteria:

* 1. History of any type of atrial fibrillation. 2. Receiving pharmacological treatments with potential impact on heart rhythm. 3. History of potentially malignant ventricular arrhythmias. 4. Uncontrolled hypothyroidism or hyperthyroidism. 5. Significant chronic obstructive pulmonary disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Hypertensive patients older than 75 years or between 65 to 75 years with moderate-high risk developing atrial fibrilation by HARMS2-AF score > 5 or a modified Taiwan AF score > 4
Sampling Method: Probability Sample
Enrollment: 499 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
new atrial fibrillation | one year
  The MODO PA/AF study will seek to determine the number of hypertensive patients who develop new atrial fibrillation, whether symptomatic or asymptomatic. As well as building an algorithm with artificial intelligence to determine the risk of suffering from a new atrial fibrillation
The absolute numbers of patients with new atrial fibrillation | one year
  The primary outcome measure of MODE BP/AF study is to detect subclinical atrial fibrillation. A central core lab is in charge of reading the ECG strips and reporting the research team new atrial fibrillation.
The percentage of patients with new atrial fibrillation | one year
  The primary outcome measure of MODE BP/AF study is to detect subclinical atrial fibrillation. A central core lab is in charge of reading the ECG strips and reporting the research team new atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Piskorz, MD, Study Chair — British Sanatorium Cardiovascular Research Center
Locations (1):
- British Sanatorium Cardiovascular Research Center, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
all database
Supporting Information: Study Protocol, SAP, CSR
Time Frame: year 2026 no end date
Access Criteria: free access. You are reporting that the URL does not appear to link to a functioning web page. But the URL is wotking
URL: http://cicbritanico.com.ar

REFERENCES:
- [Derived] Piskorz D, Lopez-Santi R, Piskorz G, Perez M, Juarez-Lloclla J, Palomo-Pinon S, Anchique-Santos C, Cardenas-Castellanos J, Nuriulu P, De Las Salas-Perez H, Ruise M, Brondello S, Del Sueldo M, Duarte-Vera Y, Munera-Echeverri A, Celis D, Miranda G, Norabuena-Rossel L, Marino M, Alvarez-Lopez H, Cedeno-Zambrano MJ, Rocha-Enciso L, Galvan-Oseguera H, Ramos-Carrillo F, Penaherrera-Oviedo M. Home monitoring for the detection of atrial fibrillation in hypertensive patients. BP/AF MODE study. Arch Cardiol Mex. 2026 Jan 12. doi: 10.24875/ACM.25000149. Online ahead of print. PMID 41525689
- See also: research center webpage. You are reporting that the URL does not appear to link to a functioning web page. But the URL is wotking — https://www.cicbritanico.com.ar/
- Available data/document: Study Protocol: British Sanatorium CIC — https://www.cicbritanico.com.ar/ — data will be at the website.You are reporting that the URL does not appear to link to a functioning web page. But the URL is wotking